CLINICAL TRIAL: NCT06976203
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of KarXT + KarX-EC for the Treatment of Cognitive Impairment Associated With Mild to Moderate Alzheimer's Disease (MINDSET 2)
Brief Title: A Study to Evaluate the Efficacy and Safety of KarXT + KarX-EC for Cognitive Impairment in Alzheimer's Disease (MINDSET 2)
Acronym: MINDSET 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN012-0052; 2025-520747-32 (Other: EU CTR); U1111-1317-4515 (Other: WHO)
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Cognitive Impairment; Kar-XT; KarX-EC; Mild Alzheimer's Disease; Moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT + KarX-EC (Active Comparator)
  Interventions: Drug: KarXT; Drug: KarX-EC
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510
  Arms: KarXT + KarX-EC
Drug: KarX-EC — Specified dose on specified days
  Other Names: BMS-986519
  Arms: KarXT + KarX-EC
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KarXT + KarX-EC for cognitive impairment in Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a confirmed diagnosis of Alzheimer's disease (AD), specifically at the mild (stage 4) or moderate (stage 5) dementia stages, as defined by the National Institute on Aging and Alzheimer's Association (NIA-AA) core clinical criteria. The diagnosis of AD pathology must be confirmed through the 2024 revised NIA-AA Workgroup criteria using a stepwise diagnostic approach.
* Participants must have an Mini-Mental State Examination (MMSE) score ranging from 12 through 22, inclusive, at the time of screening.
* Participants must have a designated caregiver who maintains adequate contact (around 10 hours per week or more) and is willing to attend all study visits. The caregiver must also be responsible for reporting on the participant's condition, overseeing medication compliance, and consenting to their involvement in both their own and the participant's study-related activities.
* Participants on acetyl choline esterase inhibitors (AChEIs) and/or memantine, must have been on a stable dosage for at least 12 weeks prior to screening, and agree to maintain this stable dose for the study duration.

Exclusion Criteria:

Participants must not present with any significant or severe medical conditions that could compromise their safety, the ability to comply with or complete the study, or the integrity of the study results. This includes any grade of hepatic impairment, urinary retention, active biliary disease, moderate-severe renal impairment (eGFR of <50 mL/min), and unstable hypertension or tachycardia.

* Participants must not have any primary psychiatric diagnoses such as major depression, schizoaffective disorder, or bipolar disorder, and those with severe psychiatric symptoms that could complicate the interpretation of treatment effects, impair cognitive assessment, or impact study completion.
* Participants must not have a history of schizophrenia or other chronic psychosis, as well as those who have previously been exposed to KarXT or are currently undergoing treatment with disease-modifying anti-amyloid therapies for AD within the past 6 months prior to screening.
* Participants must not have significant pathological findings on brain magnetic resonance imaging (MRI) at screening that could affect safety or interfere with study procedures.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2028-09-11 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Alzheimer's Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog11) | At week 24
Clinician's Interview-Based Impression Plus Caregiver Input (CIBIC+) | At week 24

SECONDARY OUTCOMES:
Change from baseline in Alzheimer's Disease Cooperative Study-Activities of Daily Living scale (ADCS-ADL) | At week 24
Change from baseline in neuro psychiatric inventory (NPI) total score | At week 24
Number of participants with adverse events (AEs) | At week 24
Number of participants with serious adverse events (SAEs) | At week 24
Number of participants with adverse event of special interest (AESIs) | At week 24
Number of participants with AEs leading to study intervention discontinuation | At week 24
Number of participants with AEs leading to study discontinuation | At week 24
Number of participants with AEs leading to death | At week 24
Number of participants with clinically significant changes in vital signs | At week 24
Number of participants with clinically significant changes in electrocardiogram (ECG) tests | At week 24
Number of participants with clinically significant changes in Columbia-Suicide Severity Rating Scale (C-SSRS) tests | At week 24
Number of participants with clinically significant changes in weight | At week 24
Number of participants with clinically significant changes in safety laboratory tests | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (120):
- United States (30):
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Inglewood Clinical, Inglewood, California
  - Irvine Clinical Research, Irvine, California
  - Local Institution - 0083, Palo Alto, California
  - Local Institution - 0069, San Diego, California
  - Local Institution - 0088, Colorado Springs, Colorado
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - K2 MEDICAL Research THE VILLAGES, Lady Lake, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Local Institution - 0080, Watertown, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Private Practice - Dr. Ronald Louis Schwartz, Hattiesburg, Mississippi
  - Local Institution - 0119, Ridgewood, New Jersey
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Clinical Institute, West Long Branch, New Jersey
  - Neurological Associates Albany, Albany, New York
  - Local Institution - 0068, Amherst, New York
  - University at Buffalo - UBMD Neurology, Buffalo, New York
  - Local Institution - 0078, Lake Success, New York
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Local Institution - 0081, Dallas, Texas
  - Central Texas Neurology Consultants, PA, Round Rock, Texas
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (6):
  - Local Institution - 0029, ABB, Buenos Aires F.D.
  - Local Institution - 0027, Córdoba, Córdoba Province
  - Local Institution - 0025, Buenos Aires
  - Local Institution - 0028, Córdoba
  - Local Institution - 0030, Córdoba
  - Local Institution - 0026, Mendoza
- Australia (4):
  - Local Institution - 0055, Saint Lucia, Queensland
  - Local Institution - 0053, Sippy Downs, Queensland
  - Griffith University - Gold Coast Campus, Southport, Queensland
  - Local Institution - 0054, Ivanhoe, Victoria
- Brazil (4):
  - Local Institution - 0115, Fortaleza, Ceará
  - Local Institution - 0101, Maringá, Paraná
  - Local Institution - 0099, Rio de Janeiro
  - Local Institution - 0100, São Paulo
- Finland (5):
  - Terveystalo Oulu, Oulu, North Ostrobothnia
  - Local Institution - 0009, Turku, Southwest Finland
  - CRST Helsinki Oy, Helsinki, Uusimaa
  - Terveystalo Ruoholahti, Helsinki
  - Itä-Suomen Yliopisto Kuopio, Kuopio
- France (12):
  - Assistance Publique Hôpitaux de Marseille - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Centre Hospitalier Universitaire Toulouse - Cité de la Santé, Toulouse, Haute-Garonne
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Roger Salengro, Lille, Hauts-de-France
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire Régional de Nancy, Nancy, Meurthe-et-Moselle
  - Hospices Civils de Lyon - Hôpital Pierre Wertheimer, Bron, Rhône
  - Local Institution - 0017, Villefranche-sur-Saône, Rhône
  - Bordeaux University Hospital - Pellegrin, Bordeaux
  - Assistance Publique Hôpitaux de Paris - Groupe Hospitalier 10e - Hôpital Lariboisière, Paris
  - Hôpital Broca, Paris
  - Pitie Salpetriere University Hospital, Paris
  - Les Hôpitaux Universitaires de Strasbourg - Hôpital de la Robertsau, Strasbourg
- Germany (6):
  - Local Institution - 0004, Munich, Bavaria
  - Local Institution - 0023, Göttingen, Lower Saxony
  - Private Practice - Dr. Irma Schöll, Bad Homburg
  - Pharmakologisches Studienzentrum Chemnitz, Chemnitz
  - Universitaetsklinikum Koeln, Cologne
  - Local Institution - 0003, Ulm
- Greece (5):
  - Local Institution - 0109, Pátrai, Achaḯa
  - University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí
  - Local Institution - 0061, Marousi, Attikí
  - Local Institution - 0059, Ioannina, Ioánnina
  - Local Institution - 0110, Thessaloniki
- Italy (3):
  - Local Institution - 0057, Napoli, Campania
  - Azienda Ospedaliero Universitaria Policlinico Riuniti di Foggia, Foggia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
- Japan (14):
  - Local Institution - 0121, Inage, Chiba
  - Local Institution - 0123, Matsudo, Chiba
  - Local Institution - 0124, Higashihiroshima, Hiroshima
  - Local Institution - 0120, Kita, Kagawa-ken
  - Kokankai Kokan Clinic, Kawasaki, Kanagawa
  - Local Institution - 0106, Kawasaki, Kanagawa
  - Local Institution - 0038, Ina, Nagano
  - National Hospital Organization Niigata Hospital, Kashiwazaki, Niigata
  - Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Local Institution - 0035, Osaka, Osaka
  - National Hospital Organization Hizen Psychiatric Center, Yoshinogari-cho, Kanzaki-gun, Saga-ken
  - Local Institution - 0037, Wako, Saitama
  - Local Institution - 0112, Wako, Saitama
  - Local Institution - 0107, Kyoto
- Netherlands (3):
  - Brain Research Center Den Bosch B.V., 's-Hertogenbosch, North Brabant
  - Brain Research Center, Amsterdam, North Holland
  - Brain Research Center Zwolle, Zwolle, Overijssel
- Poland (4):
  - Local Institution - 0066, Oświęcim, Lesser Poland Voivodeship
  - Local Institution - 0064, Wroclaw, Lower Silesian Voivodeship
  - Local Institution - 0108, Lublin, Lublin Voivodeship
  - Local Institution - 0065, Katowice, Silesian Voivodeship
- Portugal (6):
  - Campus Neurológico Sénior, Torres Vedras, Lisbon District
  - Local Institution - 0104, Matosinhos Municipality, Porto District
  - Hospital de Braga, Braga
  - Local Institution - 0049, Coimbra
  - Local Institution - 0063, Guimarães
  - Local Institution - 0052, Porto
- SCB Research Center, Bayamón, Puerto Rico
- Romania (4):
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest, București
  - Local Institution - 0113, Constanța, Constanța County
  - Local Institution - 0042, Bucharest
  - Local Institution - 0041, Sanpetru /Brasov
- Spain (7):
  - Fundació ACE, Barcelona, Barcelona [Barcelona]
  - Policlinica Gipuzkoa, Donostia / San Sebastian, Basque Country
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Doctor Peset, Valencia, Valenciana, Comunitat
  - Complejo Hospitalario Ruber Juan Bravo, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (6):
  - Local Institution - 0097, Manchester, England
  - Local Institution - 0111, Kippax, Leeds
  - Local Institution - 0116, London, London, City of
  - Local Institution - 0103, Edinburgh, Midlothian
  - Warneford Hospital, Oxford, Oxfordshire
  - Re:Cognition Health - Birmingham, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06976203.html